CLINICAL TRIAL: NCT03610594
Title: Effects of Kalaripayattu on Psychological Wellbeing and Behavior in Children: Randomised Wait- List Control Trial
Brief Title: Effects of Kalaripayattu on Psychological Wellbeing and Behavior in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NMP Medical Research Institute (Other)
Collaborators: Warwick Research Services (Other); Swamigal Trust for Vedic Science, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STVS 023
Record Dates: First submitted 2018-07-26; First posted 2018-08-01 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Psychological; Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kalaripayattu (Experimental): The experimental groups will treated with kalaripayattu exercises for the period of 12 weeks
  Interventions: Other: Kalaripayattu
- Wait list control (No Intervention): Control group will not be given any intervention. After the treatment period is over, all the subjects will be given Kalaripayattu training.

INTERVENTIONS:
Other: Kalaripayattu — Combination of Exercise, breathing, meditation, combat practices
  Arms: kalaripayattu

SUMMARY:
Kalaripayattu is an ancient martial art of India which has been practiced for centuries. It is mentioned in Vedic litrature of Ayurveda,Dhanurveda and Yoga. The main elements of Kalaripayattu include training in physical, combat, breathing exercises, higher form of meditation and specific class of medical treatments. The purpose of the experimental study is to determine the effect of kalaripayattu on psychological well-being and behaviour in children.

ELIGIBILITY:
Inclusion Criteria:

* Children from 8 years to 12 years of age
* Parents agreed to informed consent

Exclusion Criteria:

* Physical disabilities
* Diagnosed Mental or behavioural disorder
* Practicing other exercise, physical trainings or yoga

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Psychological Well-being | Change from baseline to 12 weeks
  Measured by MacArthur Health and Behavior Questionnaire

SECONDARY OUTCOMES:
Behavior | Change from baseline to 12 weeks
  Measured by Child Behavior Scale

CONTACTS AND LOCATIONS:
Overall Officials: Neha sharma, PhD, Study Director — Warwick Research Services; Ravishankar Ramanathan, BA, Principal Investigator — Swamigal Trust for Vedic Studies
Locations (1):
- NMP Medical Reserach Institute, Jaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: Undecided